CLINICAL TRIAL: NCT03864068
Title: Inositol Supplementation to Treat Polycystic Ovary Syndrome: A Double Blind Dose Ranging RCT (INSUPP-PCOS)
Brief Title: Inositol Supplementation to Treat PCOS (INSUPP-PCOS)
Acronym: INSUPP-PCOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Richard S. Legro, M.D., Chair, Obstetrics and Gynecology, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Study00010252; 1R01AT009484-01A1 (NIH)
Record Dates: First submitted 2019-03-04; First posted 2019-03-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Polycystic Ovary Syndrome; Anovulation; Hyperandrogenism; Insulin Resistance; Glucose Intolerance; Metabolic Complication
Keywords: Polycystic Ovary Syndrome; Anovulation; Hyperandrogenism; Insulin Resistance; Glucose Intolerance; Metabolic Complication
MeSH Terms: conditions — Polycystic Ovary Syndrome; Anovulation; Hyperandrogenism; Insulin Resistance; Glucose Intolerance | interventions — maltodextrin; Inulin; Inositol

STUDY DESIGN:
Intervention Model Description: Placebo Group; Active Treatment with Inositol 1gm/bid; Active Treatment with Inositol 2gm/bid; Active Treatment with Inositol 3gm/ bid
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo Treatment bid (Placebo Comparator): Women with PCOS (N = 30) will receive the daily placebo (maltodextrin and inulin) in an identical fashion as the active study group and will be monitored the same.
  Interventions: Other: Placebo
- Active Treatment with Inositol 1gm/bid (Experimental): Women with PCOS (N = 30) will receive daily inositol powder BID as active drug (each dose with 1000 mg of myo-inositol and 25 mg of d-chiro-inositol) over the initial 3 mos RCT period.
  Interventions: Drug: Inositol
- Active Treatment with Inositol 2 gm/bid (Experimental): Women with PCOS (N = 30) will receive daily inositol powder BID as active drug (each dose with 2000 mg of myo-inositol and 50 mg of d-chiro-inositol) over the initial 3 mos RCT period.
  Interventions: Drug: Inositol
- Active Treatment with Inositol 3 gm/bid (Experimental): Women with PCOS (N = 30) will receive daily inositol powder BID as active drug (each dose with 3000 mg of myo-inositol and 75 mg of d-chiro-inositol) over the initial 3 mos RCT period.
  Interventions: Drug: Inositol

INTERVENTIONS:
Other: Placebo — Placebo
  Other Names: maltodextrin and inulin
  Arms: Placebo Treatment bid
Drug: Inositol — 1gm/bid, 2gm/bid or 3gm/bid of Inositol powder
  Arms: Active Treatment with Inositol 1gm/bid; Active Treatment with Inositol 2 gm/bid; Active Treatment with Inositol 3 gm/bid

SUMMARY:
To determine if Inositol, a dietary supplement, will improve ovarian and adrenal androgen excess in women with Polycystic Ovarian Syndrome(PCOS).

DETAILED DESCRIPTION:
This trial will test prospectively the effects of inositol supplementation in a dose ranging double blind randomized controlled trial, according to CONSORT guidelines. This will be a four armed study of three doses of inositol vs. placebo over a three month period with the reduction in hyperandrogenism (based on serum testosterone levels) as the primary outcome and key secondary outcomes of the change in sex hormone binding globulin(SHBG) and the related free androgen index, fasting insulin levels and area under the curve glucose levels from an oral glucose challenge test (OGTT). The hypothesis is that women with PCOS who receive inositol supplementation will have a dose related reduction in hyperandrogenism. Further, we propose that the primary mechanism of inositol will be a significant improvement in hyperandrogenism (both ovarian and adrenal) vs. placebo, as documented by a lower free androgen index [decreased total testosterone and increased sex hormone blinding globulin (SHBG)], lower sebum measures and lower antral follicle counts of the ovary and anti-Mullerian hormone, all of which will correlate with the decrease in hyperandrogenism.

ELIGIBILITY:
Inclusion Criteria:

* Women with chronic anovulation or oligomenorrhea defined as spontaneous intermenstrual periods of greater than or equal to 45 days or a total of less than or equal to 8 menses per year.
* Women with Hyperandrogenism defined as a total testosterone greater than 50 ng/dL or a free androgen index greater than 10.
* Women with Polycystic Ovaries on Ultrasound defined as either 12 or more follicles measuring 2-9 mm in diameter or increased ovarian volume greater than 10 cm.

Exclusion Criteria:

* Women with Hyperprolactinemia defined as 2 prolactin levels at least one week apart greater than 30 ng/mL.
* Women with known 21-hydroxylase deficiency or other enzyme deficiency leading to the congenital adrenal hyperplasia.
* Women with elevated FSH levels greater than 10 mIU/mL.
* Women with uncorrected thyroid disease as per ASRM guidelines for nonpregnant subjects (TSH less than 0.45 mIU/mL or greater than 4.5 MIU/mL).
* Women with a suspected adrenal or ovarian tumor secreting androgens
* Women with Cushing's syndrome
* Women on confounding medications which affect ovarian function including metformin, hormonal contraceptives or other medications for type 2 diabetes
* Women with medical conditions that are contraindications to OTC inositol or previous allergic reactions to the supplement or to the placebo maltodextrin or inulin.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — PCOS is a disorder that only affects women and therefore men are not eligible to participate in this study.
Enrollment: 154 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Change in total testosterone | baseline and 3 months
  Serum total testosterone levels

SECONDARY OUTCOMES:
Change in SHBG | baseline and 3 months
  SHBG levels
Change in Free Androgen Index (FAI) | baseline and 3 months
  FAI levels
Change in area under the curve (AUC) of glucose | baseline and 3 months
  AUC of a 2-hour 75g glucose tolerance test, which measures glucose at 0, 30, 60, 90, and 120 minutes.
Change in fasting insulin | baseline and 3 months
  Fasting insulin levels

CONTACTS AND LOCATIONS:
Overall Officials: Richard S. Legro, M.D., Principal Investigator — Penn State College of Medicine, Hershey Medical Center
Locations (2):
- United States (2):
  - Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania